CLINICAL TRIAL: NCT00689728
Title: A Phase 2 Study of Multiple Intravenous Doses of LY2127399 in Patients With Rheumatoid Arthritis on Concomitant Methotrexate and an Inadequate Response to TNFα Inhibitor Therapy
Brief Title: A Study for Patients With Rheumatoid Arthritis on Methotrexate (MTX) With an Inadequate Response to TNFα Inhibitor Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11351; H9B-MC-BCDG (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Results first posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-11

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tabalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 30 milligram (mg) LY2127399 (Experimental): Double-blind Treatment: 30 mg LY2127399 administered as a single intravenous (IV) infusion over 30 minutes at 0, 3, and 6 weeks.
  Rescue: At Week 16 primary endpoint, participants without at least 20% improvement in either tender or swollen joint counts based on 28 joints, could receive an additional (unblinded) 30 minute infusion of LY2127399 80 mg or remain on initial randomized treatment up to Week 24.
  Follow-up: Optional visits beyond Week 24, if needed, to assess safety including B cell count recovery.
  Interventions: Biological: LY2127399
- 80 mg LY2127399 (Experimental): Double-blind Treatment: 80 mg LY2127399 administered as a single IV infusion over 30 minutes at 0, 3, and 6 weeks.
  Rescue: At Week 16 primary endpoint, participants without at least 20% improvement in either tender or swollen joint counts based on 28 joints, could receive an additional (unblinded) 30 minute infusion of LY2127399 80 mg or remain on initial randomized treatment up to Week 24.
  Follow-up: Optional visits beyond Week 24, if needed, to assess safety including B cell count recovery.
  Interventions: Biological: LY2127399
- Placebo (Placebo Comparator): Double-blind Treatment: Placebo comparator administered as a single IV infusion over 30 minutes at 0, 3, and 6 weeks.
  Rescue: At Week 16 primary endpoint, participants without at least 20% improvement in either tender or swollen joint counts based on 28 joints could receive an additional (unblinded) 30 minute infusion of LY2127399 80 mg or remain on same initial randomized treatment up to Week 24.
  Follow-Up: Optional visits beyond Week 24, if needed, to assess safety including B cell count recovery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: LY2127399 — LY2127399 will be administered as a single IV infusion over 30 minutes.
  Arms: 30 milligram (mg) LY2127399; 80 mg LY2127399
Drug: Placebo — Placebo will be administered as a single IV infusion over 30 minutes.
  Arms: Placebo

SUMMARY:
The purpose of this study is to explore whether LY2127399 is effective in relieving signs and symptoms of rheumatoid arthritis (RA) in patients with a history of inadequate response or intolerance to at least 1 Tumor Necrosis Factor-Alpha (TNFα) inhibitor therapy. Examples of these TNFα inhibitor therapies that are currently on the market include Enbrel® (etanercept), Remicade® (infliximab), and Humira® (adalimumab).

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent approval
* Women must not be at risk to become pregnant during study participation
* Diagnosis of Rheumatoid Arthritis
* Active Rheumatoid Arthritis
* Current, regular use of Methotrexate, at a stable dose
* Have been on at least 1 biologic tumor necrosis factor-alpha (TNFα) inhibitor therapy and either failed or were intolerant to treatment
* Other criteria to be reviewed by study doctor

Exclusion Criteria:

* Use of excluded medications (reviewed by study doctor)
* Have medical findings which, in the opinion of the study doctor, put patient at an unacceptable risk for participation in the study
* Have had recent or ongoing infection which, in the opinion of the study doctor put patient at an unacceptable risk for participation
* Evidence of tuberculosis
* Have systemic inflammatory condition other than rheumatoid arthritis (RA), such as juvenile RA, seronegative spondyloarthropathy, Crohn's disease, ulcerative colitis, or psoriatic arthritis.
* Other criteria to be reviewed by study doctor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-06; Primary Completion 2010-02 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (45):
- United States (19):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mesa, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palm Desert, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Riverside, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Maria, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Upland, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jupiter, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vero Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zephyrhills, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hickory, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Middleburg Heights, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orangeburg, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mesquite, Texas
- Argentina (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Miguel de Tucumán
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna, Austria
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liège, Belgium
- Brazil (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Campinas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Curitiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goiânia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto Alegre
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Setor Oeste/Goiania
- Canada (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamilton, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kitchener, Ontario
- Germany (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Göttingen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hildesheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vogelsang
- Mexico (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chihuahua City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cuernavaca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morelia
- Poland (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan, Puerto Rico

REFERENCES:
- [Derived] Genovese MC, Fleischmann RM, Greenwald M, Satterwhite J, Veenhuizen M, Xie L, Berclaz PY, Myers S, Benichou O. Tabalumab, an anti-BAFF monoclonal antibody, in patients with active rheumatoid arthritis with an inadequate response to TNF inhibitors. Ann Rheum Dis. 2013 Sep 1;72(9):1461-8. doi: 10.1136/annrheumdis-2012-202775. Epub 2012 Dec 25. PMID 23268367
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Double-blind treatment was administered at Weeks 0, 3, and 6. At Week 16, participants not having at least a 20% decrease in tender or swollen joint counts could receive rescue therapy. Post-study B-cell follow-up (safety only) occurred beyond Week 24.
Groups:
- 30 mg LY2127399: Double-blind: 30 mg LY2127399 administered as a single intravenous (IV) infusion over 30 minutes at 0, 3, and 6 weeks.
  Rescue: either remain on 30 mg LY2127399 or receive 80 mg LY2127399 up to Week 24.
  Optional Follow-up: assessing safety after Week 24, if needed.
- 80 mg LY2127399: Double-blind: 80 mg LY2127399 administered as a single intravenous (IV) infusion over 30 minutes at 0, 3, and 6 weeks.
  Rescue: remain on 80 mg LY2127399 up to Week 24. Optional Follow-up: assessing safety after Week 24, if needed.
- Placebo: Double-blind: Placebo comparator administered as a single intravenous (IV) infusion over 30 minutes at 0, 3, and 6 weeks.
  Rescue: either remain on placebo or receive 80 mg LY2127399 up to Week 24. Optional Follow-up: assessing safety after Week 24, if needed.
Period: Double-Blind Treatment
Arm/Group | 30 mg LY2127399 | 80 mg LY2127399 | Placebo
Started | 35 | 30 | 35
Completed | 31 | 26 | 30
Not Completed | 4 | 4 | 5
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 3 | 2
Not completed — Lack of Efficacy | 0 | 1 | 2
Period: Rescue
Arm/Group | 30 mg LY2127399 | 80 mg LY2127399 | Placebo
Started | 31 | 26 | 30
Completed | 30 | 24 | 29
Not Completed | 1 | 2 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1
Period: Optional Follow-Up
Arm/Group | 30 mg LY2127399 | 80 mg LY2127399 | Placebo
Started | 9 (21 participants who completed the rescue period did not enter the optional follow-up period.) | 11 (13 participants who completed the rescue period did not enter the optional follow-up period.) | 10 (19 participants who completed the rescue period did not enter the optional follow-up period.)
Completed | 6 | 5 | 4
Not Completed | 3 | 6 | 6
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- 30 mg LY2127399: 30 mg LY2127399 administered as a single intravenous (IV) infusion over 30 minutes at 0, 3, and 6 weeks.
- 80 mg LY2127399: 80 mg LY2127399 administered as a single intravenous (IV) infusion over 30 minutes at 0, 3, and 6 weeks.
- Placebo: Placebo comparator administered as a single intravenous (IV) infusion over 30 minutes at 0, 3, and 6 weeks.
- Total: Total of all reporting groups
Arm/Group | 30 mg LY2127399 | 80 mg LY2127399 | Placebo | Total
Number analyzed (Participants) | 35 | 30 | 35 | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.4 (13.03) | 52.7 (14.05) | 52.2 (11.46) | 52.4 (12.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 26 | 32 | 86
  Male | 7 | 4 | 3 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 26 | 20 | 21 | 67
  African | 3 | 3 | 8 | 14
  Hispanic | 6 | 7 | 6 | 19
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 18 | 14 | 50
  Puerto Rico | 0 | 0 | 1 | 1
  Canada | 2 | 1 | 1 | 4
  Argentina | 4 | 4 | 4 | 12
  Poland | 1 | 1 | 4 | 6
  Belgium | 0 | 1 | 0 | 1
  Brazil | 6 | 3 | 6 | 15
  Austria | 2 | 2 | 3 | 7
  Germany | 2 | 0 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology (ACR)50 Response at Week 16
Description: ACR50 Responder Index is a composite of clinical, laboratory, and functional measures in rheumatoid arthritis. ACR50 Responder is defined as a participant with greater than 50% improvement from baseline in both tender and swollen joint counts and in at least 3 of the following 5 criteria: physician global assessment, patient global assessment, functional ability measure (Health Assessment Questionnaire-Disability Index which measures participants' perceived degree of difficulty when performing various daily activities), visual analog pain scale, and erythrocyte sedimentation rate or C-reactive protein.
Time Frame: 16 weeks
Population: Non-responder imputation/last observation carried forward (NRI/LOCF); intention to treat (ITT) population defined as participants who were randomized, received at least one dose of study drug, and had at least one post-baseline ACR50 assessment. Two participants from sites with good clinical practice [GCP] violations are excluded.
Measure: Number; unit: Percentage of Participants
Arm/Group | 30 mg LY2127399 | 80 mg LY2127399 | Placebo
Number analyzed (Participants) | 35 | 28 | 35
Percentage of Participants | 11.4 | 14.3 | 2.9
Statistical Analysis 1: Comparison: 30 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.178, Fisher Exact
Statistical Analysis 2: Comparison: 80 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.116, Fisher Exact

2. Secondary Outcome: Number of Participants Experiencing An Adverse Event
Description: Serious adverse events and other non-serious adverse events are located in the Reported Adverse Event section.
Time Frame: Baseline up to 68 weeks
Population: Safety population defined as all participants who were randomized and received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- 30 mg LY2127399 - Treatment; 30 mg LY2127399 - Without Rescue Treatment: 30 mg LY2127399 administered as a single intravenous (IV) infusion over 30 minutes at 0, 3, and 6 weeks.
- 80 mg LY2127399 - Treatment; 80 mg LY2127399 - Without Rescue Treatment: 80 mg LY2127399 administered as a single intravenous (IV) infusion over 30 minutes at 0, 3, and 6 weeks.
- Placebo - Treatment; Placebo - Without Rescue Treatment: Placebo comparator administered as a single intravenous (IV) infusion over 30 minutes at 0, 3, and 6 weeks.
- 30 mg LY2127399 - With Rescue Treatment: Participants who were randomized to LY2127399 30 mg during Treatment Phase who did not have an improvement of at least 20% in either their tender or their swollen joint counts, based on 28 joints at Week 16 assessments and chose to receive optional rescue treatment of an additional 30 minute infusion of LY2127399 80 mg at Week 16.
- 80 mg LY2127399 - With Rescue Treatment: Participants who were randomized to LY2127399 80 mg during Treatment Phase who did not have an improvement of at least 20% in either their tender or their swollen joint counts, based on 28 joints at Week 16 assessments and chose to receive optional rescue treatment of an additional 30 minute infusion of LY2127399 80 mg at Week 16.
- Placebo - With Rescue Treatment: Participants who were randomized to placebo during Treatment Phase who did not have an improvement of at least 20% in either their tender or their swollen joint counts, based on 28 joints at Week 16 assessments and chose to receive optional rescue treatment of an additional 30 minute infusion of LY2127399 80 mg at Week 16.
- 30 mg LY2127399 - Follow Up: Participants who were randomized to LY2127399 30 mg during Treatment Phase who required additional follow-up for monitoring of their B cell counts, regardless of whether or not they received optional rescue treatment of an additional 30 minute infusion of LY2127399 80 mg at Week 16.
- 80 mg LY2127399 - Follow Up: Participants who were randomized to LY2127399 80 mg during Treatment Phase who required additional follow-up for monitoring of their B cell counts, regardless of whether or not they received optional rescue treatment of an additional 30 minute infusion of LY2127399 80 mg at Week 16.
- Placebo - Follow Up: Participants who were randomized to placebo during Treatment Phase who required additional follow-up for monitoring of their B cell counts, regardless of whether or not they received optional rescue treatment of an additional 30 minute infusion of LY2127399 80 mg at Week 16.
Arm/Group | 30 mg LY2127399 - Treatment | 80 mg LY2127399 - Treatment | Placebo - Treatment | 30 mg LY2127399 - Without Rescue Treatment | 30 mg LY2127399 - With Rescue Treatment | 80 mg LY2127399 - Without Rescue Treatment | 80 mg LY2127399 - With Rescue Treatment | Placebo - Without Rescue Treatment | Placebo - With Rescue Treatment | 30 mg LY2127399 - Follow Up | 80 mg LY2127399 - Follow Up | Placebo - Follow Up
Number analyzed (Participants) | 35 | 30 | 35 | 19 | 12 | 15 | 11 | 10 | 20 | 9 | 11 | 10
Participants
  Serious | 1 | 2 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other | 22 | 21 | 22 | 2 | 5 | 6 | 3 | 3 | 11 | 1 | 4 | 1

3. Secondary Outcome: Change From Baseline in Medical Outcome Study 36-Item Short Form Health Survey (SF-36) at Week 16
Description: Self-reported questionnaire of 36 questions in 8 domains (physical functioning, social functioning, bodily pain, vitality, mental health, role-physical, role-emotional, general health). Each domain is scored by summing individual items and transforming scores into a 0-100 scale (higher scores=better health status/function). The mental and physical component summaries are based on the 8 domains. Component scores are transformed scores representing a mean (50) and standard deviation (10) in the general United States (US) population. Scores > or <50 are above or below the average US population.
Time Frame: Baseline, 16 weeks
Population: Intention to treat (ITT) population defined as participants who were randomized, received at least one dose of study drug, and had at least one post-baseline SF-36 assessment; last observation carried forward (LOCF). Two participants from sites with good clinical practice [GCP] violations are excluded.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | 30 mg LY2127399 | 80 mg LY2127399 | Placebo
Number analyzed (Participants) | 34 | 27 | 34
Units on a Scale
  Physical Health | 5.064 (8.73) | 5.197 (8.36) | 1.229 (6.18)
  Mental Health | 2.700 (10.82) | 3.597 (11.96) | 0.133 (12.99)
Statistical Analysis 1: Comparison: 30 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.062, ANCOVA — p-value represents change from baseline at 16 weeks for LY2127399 30 mg. vs. placebo in Physical Health Component scores; Mean Difference (Final Values) = 4.873
Statistical Analysis 2: Comparison: 80 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.052, ANCOVA — p-value represents change from baseline at 16 weeks for LY2127399 80 mg. vs. placebo in Physical Health Component scores; Mean Difference (Final Values) = 5.427
Statistical Analysis 3: Comparison: 30 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.655, ANCOVA — p-value represents change from baseline at 16 weeks for LY2127399 30 mg. vs. placebo in Mental Health Component scores; Mean Difference (Final Values) = 1.720
Statistical Analysis 4: Comparison: 80 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.173, ANCOVA — p-value represents change from baseline at 16 weeks for LY2127399 80 mg. vs. placebo in Mental Health Component scores; Mean Difference (Final Values) = 4.264

4. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology (ACR) 20 Response at Week 16
Description: ACR20 Responder Index is a composite of clinical, laboratory, and functional measures in rheumatoid arthritis. An ACR20 Responder is defined as a participant with at least 20% improvement from baseline in both tender and swollen joint counts and in at least 3 of the following 5 criteria: physician global assessment, patient global assessment, functional ability measure (Health Assessment Questionnaire-Disability Index which measures participants' perceived degree of difficulty when performing various daily activities), visual analog pain scale, and erythrocyte sedimentation rate or C-reactive protein.
Time Frame: 16 weeks
Population: Non-responder imputation (NRI)/last observation carried forward; intention to treat (ITT) population defined as participants who were randomized, received at least one dose of study drug, and had at least one post-baseline ACR20 assessment. Two participants from sites with good clinical practice [GCP] violations are excluded.
Measure: Number; unit: Percentage of Participants
Arm/Group | 30 mg LY2127399 | 80 mg LY2127399 | Placebo
Number analyzed (Participants) | 35 | 28 | 35
Percentage of Participants | 25.7 | 28.6 | 17.1
Statistical Analysis 1: Comparison: 30 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.281, Fisher Exact
Statistical Analysis 2: Comparison: 80 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.218, Fisher Exact

5. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology (ACR)70 Response at Week 16
Description: ACR70 Responder Index is a composite of clinical, laboratory, and functional measures in rheumatoid arthritis. An ACR70 Responder is defined as a participant with at least 70% improvement from baseline in both tender and swollen joint counts and in at least 3 of the following 5 criteria: physician global assessment, patient global assessment, functional ability measure (Health Assessment Questionnaire-Disability Index which measures participants' perceived degree of difficulty when performing various daily activities), visual analog pain scale, and erythrocyte sedimentation rate or C-reactive protein.
Time Frame: 16 weeks
Population: Non-responder imputation (NRI)/last observation carried forward; intention to treat (ITT) population defined as participants who were randomized, received at least one dose of study drug, and had at least one post-baseline ACR70 assessment. Two participants from sites with good clinical practice [GCP] violations are excluded.
Measure: Number; unit: Percentage of Participants
Arm/Group | 30 mg LY2127399 | 80 mg LY2127399 | Placebo
Number analyzed (Participants) | 35 | 28 | 35
Percentage of Participants | 2.9 | 3.6 | 0
Statistical Analysis 1: Comparison: 30 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.500, Fisher Exact
Statistical Analysis 2: Comparison: 80 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.444, Fisher Exact

6. Secondary Outcome: Change From Baseline in Tender Joint Count at Week 16
Description: The number of tender and painful joints is determined by examination of 28 joints (14 on each side) which include: the 2 shoulders, the 2 elbows, the 2 wrists, the 10 metacarpophalangeal joints, the 2 interphalangeal joints of the thumb, the 8 proximal interphalangeal joints, and the 2 knees. The joints are assessed and classified as tender or not tender.
Time Frame: Baseline, 16 weeks
Population: Intention to treat (ITT) population defined as participants who were randomized, received at least one dose of study drug, and had at least one post-baseline tender joint assessment; last observation carried forward (LOCF). Two participants from sites with good clinical practice [GCP] violations are excluded.
Measure: Mean (Standard Deviation); unit: Tender Joints
Arm/Group | 30 mg LY2127399 | 80 mg LY2127399 | Placebo
Number analyzed (Participants) | 35 | 28 | 35
Tender Joints | -4.5 (6.74) | -6.3 (4.96) | -3.3 (8.20)
Statistical Analysis 1: Comparison: 30 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.337, ANCOVA; Mean Difference (Final Values) = -4.5
Statistical Analysis 2: Comparison: 80 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.038, ANCOVA; Mean Difference (Final Values) = -6.6

7. Secondary Outcome: Change From Baseline in Swollen Joint Count at Week 16
Description: The number of swollen joints is determined by examination of 28 joints (14 on each side) which include: the 2 shoulders, the 2 elbows, the 2 wrists, the 10 metacarpophalangeal joints, the 2 interphalangeal joints of the thumb, the 8 proximal interphalangeal joints, and the 2 knees. The joints are assessed and classified as swollen or not swollen.
Time Frame: Baseline, 16 weeks
Population: Intention to treat (ITT) population defined as participants who were randomized, received at least one dose of study drug, and had at least one post-baseline swollen joint assessment; last observation carried forward (LOCF). Two participants from sites with good clinical practice [GCP] violations are excluded.
Measure: Mean (Standard Deviation); unit: Swollen Joints
Arm/Group | 30 mg LY2127399 | 80 mg LY2127399 | Placebo
Number analyzed (Participants) | 35 | 28 | 35
Swollen Joints | -2.6 (5.23) | -4.7 (4.44) | -2.3 (5.54)
Statistical Analysis 1: Comparison: 30 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.403, ANCOVA; Mean Difference (Final Values) = -2.7
Statistical Analysis 2: Comparison: 80 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.006, ANCOVA; Mean Difference (Final Values) = -5.3

8. Secondary Outcome: Change From Baseline in Participant's Assessment of Joint Pain at Week 16
Description: Participant's assessment of joint pain using a visual analog scale (VAS), which ranged from 0 to 100 millimeters, where 0 indicated no pain and 100 indicated worst possible pain.
Time Frame: Baseline, 16 weeks
Population: Intention to treat (ITT) population defined as participants who were randomized, received at least one dose of study drug, and had at least one post-baseline joint pain assessment; last observation carried forward (LOCF). Two participants from sites with good clinical practice [GCP] violations are excluded.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | 30 mg LY2127399 | 80 mg LY2127399 | Placebo
Number analyzed (Participants) | 35 | 28 | 35
Millimeters | -16.1 (26.86) | -17.8 (27.10) | -9.1 (29.20)
Statistical Analysis 1: Comparison: 30 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.168, ANCOVA; Mean Difference (Final Values) = -16.2
Statistical Analysis 2: Comparison: 80 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.075, ANCOVA; Mean Difference (Final Values) = -19.3

9. Secondary Outcome: Change From Baseline in Participant's Assessment of Disease Activity at Week 16
Description: Participant's assessment of their current arthritis disease activity using a visual analog scale (VAS), which ranged from 0 to 100 millimeters, where 0 indicated no arthritis activity and 100 indicated extremely active arthritis.
Time Frame: Baseline, 16 weeks
Population: Intention to treat (ITT) population defined as participants who were randomized, received at least one dose of study drug, and had at least one post-baseline disease activity assessment; last observation carried forward (LOCF). Two participants from sites with good clinical practice [GCP] violations are excluded.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | 30 mg LY2127399 | 80 mg LY2127399 | Placebo
Number analyzed (Participants) | 35 | 26 | 35
Millimeters | -20.2 (25.87) | -23.6 (29.36) | -11.2 (29.05)
Statistical Analysis 1: Comparison: 30 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.157, ANCOVA; Mean Difference (Final Values) = -19.3
Statistical Analysis 2: Comparison: 80 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.025, ANCOVA; Mean Difference (Final Values) = -25.6

10. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity at Week 16
Description: Physician's global assessment of arthritis disease activity using a visual analog scale (VAS) which ranged from 0 to 100 millimeters, where 0 indicates no arthritis activity and 100 indicates extremely active arthritis.
Time Frame: Baseline, 16 weeks
Population: Intention to treat (ITT) population defined as participants who were randomized, received at least one dose of study drug, and had at least one post-baseline physician's disease activity assessment; last observation carried forward (LOCF). Two participants from sites with good clinical practice [GCP] violations are excluded.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | 30 mg LY2127399 | 80 mg LY2127399 | Placebo
Number analyzed (Participants) | 35 | 27 | 35
Millimeters | -17.7 (22.55) | -17.3 (29.67) | -13.1 (26.40)
Statistical Analysis 1: Comparison: 30 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.110, ANCOVA; Mean Difference (Final Values) = -19.4
Statistical Analysis 2: Comparison: 80 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.147, ANCOVA; Mean Difference (Final Values) = -19.1

11. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) at Week 16
Description: The HAQ-DI questionnaire scores the participant's self-perception on the degree of difficulty when dressing and grooming, arising, eating, walking, hygiene, reach, grip, and performing other daily activities (0=without any difficulty, 1=with some difficulty, 2=with much difficulty, and 3=unable to do). The scores for each of the functional areas, which have a range from 0 to 3, are averaged to calculate the functional disability index. Higher scores are associated with greater disability.
Time Frame: Baseline, 16 weeks
Population: Intention to treat (ITT) population defined as participants who were randomized, received at least one dose of study drug, and had at least one post-baseline HAQ-DI assessment; last observation carried forward (LOCF). Two participants from sites with good clinical practice [GCP] violations are excluded.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | 30 mg LY2127399 | 80 mg LY2127399 | Placebo
Number analyzed (Participants) | 35 | 28 | 35
Units on a Scale | -0.161 (0.569) | -0.259 (0.623) | -0.205 (0.511)
Statistical Analysis 1: Comparison: 30 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.969, ANCOVA; Mean Difference (Final Values) = -0.172
Statistical Analysis 2: Comparison: 80 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.452, ANCOVA; Mean Difference (Final Values) = -0.280

12. Secondary Outcome: Percent Change From Baseline in C-reactive Protein (CRP) at Week 16
Time Frame: Baseline, 16 weeks
Population: Intention to treat (ITT) population defined as participants who were randomized, received at least one dose of study drug, and had at least one post-baseline CRP assessment; last observation carried forward (LOCF). Two participants from sites with good clinical practice [GCP] violations are excluded.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | 30 mg LY2127399 | 80 mg LY2127399 | Placebo
Number analyzed (Participants) | 35 | 27 | 35
Percent Change | 58.88 (216.005) | 15.14 (123.625) | 71.64 (410.942)
Statistical Analysis 1: Comparison: 30 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.554, ANCOVA
Statistical Analysis 2: Comparison: 80 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.920, ANCOVA

13. Secondary Outcome: Change From Baseline in Disease Activity Score (DAS28) at Week 16
Description: Disease Activity Score (modified to include the 28 joint count [DAS28]) consists of a composite score of the following variables: tender joint count (TJC28), swollen joint count (SJC28), C-reactive protein (CRP), and participant global assessment of their disease activity (patient global VAS). It is calculated by using the following formula:DAS28-CRP=0.56 times the square root of(28TJC)+0.28 times the square root of(28SJC)+0.36*natural log (ln)(CRP+1)+0.014*patient global VAS+0.96. Scores ranged from 1.0-9.4, where lower scores indicated less disease activity, and remission was DAS28-CRP <2.6. A decrease in DAS28-CRP indicated an improvement in participant's condition.
Time Frame: Baseline, 16 weeks
Population: Intention to treat (ITT) population defined as participants who were randomized, received at least one dose of study drug, and had at least one post-baseline DAS28 assessment; last observation carried forward (LOCF). Two participants from sites with good clinical practice [GCP] violations are excluded.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | 30 mg LY2127399 | 80 mg LY2127399 | Placebo
Number analyzed (Participants) | 35 | 26 | 34
Units on a Scale | -0.911 (1.137) | -1.288 (0.934) | -0.613 (1.041)
Statistical Analysis 1: Comparison: 30 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.100, ANCOVA; Mean Difference (Final Values) = -0.912
Statistical Analysis 2: Comparison: 80 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.005, ANCOVA; Mean Difference (Final Values) = -1.322

14. Secondary Outcome: Number of Participants With Response (Response Rate) Based Upon European League Against Rheumatism Responder Index, 28 Joint Count (EULAR28) at Week 16
Description: EULAR28 categorizes clinical response based upon improvement since baseline in Disease Activity Score modified to include the 28 joint count (DAS28) and post-baseline DAS28. DAS28 consists of a composite score of the following variables: tender joint count (TJC28), swollen joint count (SJC28), C-reactive protein (CRP), and participant global assessment of their disease activity (patient global VAS). EULAR28 categories include: No Response (improvement in DAS28 of less than or equal to 0.6 units or post-baseline DAS28 score greater than 5.1 with improvement by less than or equal to 1.2 units), Moderate Response (post-baseline DAS28 score less than or equal to 5.1 with improvement by more than 0.6 units but no greater than 1.2 units or post-baseline DAS28 score greater than 3.2 with improvement by more than 1.2 units), and Good Response (post-baseline DAS28 score less than or equal to 3.2 with improvement by more than 1.2 units).
Time Frame: 16 weeks
Population: Intention to treat (ITT) population defined as participants who were randomized, received at least one dose of study drug, and had at least one post-baseline EULAR28 assessment; last observation carried forward (LOCF). Two participants from sites with good clinical practice [GCP] violations are excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | 30 mg LY2127399 | 80 mg LY2127399 | Placebo
Number analyzed (Participants) | 35 | 26 | 34
Participants
  Good response | 5 | 5 | 0
  Moderate response | 8 | 12 | 15
  No response | 22 | 9 | 19
Statistical Analysis 1: Comparison: 30 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.022, Fisher Exact — p-value represents comparison of LY2127399-30 mg dose versus placebo for the 3 levels of EULAR response (good response, moderate response, no response)
Statistical Analysis 2: Comparison: 80 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.016, Fisher Exact — p-value represents comparison of LY2127399-80 mg dose versus placebo for the 3 levels of EULAR response (good response, moderate response, no response)

15. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Score at Week 16
Description: The FACIT Fatigue Score is a brief patient-reported measure of fatigue and consists of 13 items. Scores range from 0 to 52, with higher scores indicating less fatigue.
Time Frame: Baseline, 16 weeks
Population: Intention to treat (ITT) population defined as participants who were randomized, received at least one dose of study drug, and had at least one post-baseline FACIT assessment; last observation carried forward (LOCF). Two participants from sites with good clinical practice [GCP] violations are excluded.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | 30 mg LY2127399 | 80 mg LY2127399 | Placebo
Number analyzed (Participants) | 34 | 27 | 34
Units on a Scale | 2.5 (11.20) | 7.9 (8.44) | 3.1 (9.56)
Statistical Analysis 1: Comparison: 30 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.818, ANCOVA; Mean Difference (Final Values) = 2.6
Statistical Analysis 2: Comparison: 80 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.066, ANCOVA; Mean Difference (Final Values) = 7.7

16. Secondary Outcome: Pharmacodynamics: Change From Baseline in Absolute CD20 + B Cell Count at Week 16
Description: B-lymphocyte antigen CD20 or CD20 is an activated-glycosylated phosphoprotein expressed on the surface of all mature B-cells. For this endpoint, total B cell counts (CD20+CD3- cells) are represented by number of cells per microliter. The reference range for the absolute counts is 43-602 cells per microliter.
Time Frame: Baseline, 16 weeks
Population: Intention to treat (ITT) population defined as participants who were randomized, received at least one dose of study drug, and had at least one post-baseline CD20 assessment; last observation carried forward (LOCF). Two participants from sites with good clinical practice [GCP] violations are excluded.
Measure: Mean (Standard Deviation); unit: Cells per Microliter
Arm/Group | 30 mg LY2127399 | 80 mg LY2127399 | Placebo
Number analyzed (Participants) | 32 | 26 | 33
Cells per Microliter | -30.94 (152.813) | -34.92 (82.090) | 0.79 (144.251)
Statistical Analysis 1: Comparison: 30 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.010, ANCOVA
Statistical Analysis 2: Comparison: 80 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.056, ANCOVA

17. Secondary Outcome: Pharmacodynamics: Change From Baseline in Total B Cells (CD20 + CD3-) as a Percentage of Total Lymphocytes
Description: B-lymphocyte antigen CD20 or CD20 is an activated-glycosylated phosphoprotein expressed on the surface of all mature B-cells. For this outcome, total B cells (CD20+CD3- cells) are expressed as the relative percent of lymphocytes. There is no reference range provided for this parameter by the performing laboratory.
Time Frame: Baseline, 16 weeks
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Percentage of Lymphocytes
Arm/Group | 30 mg LY2127399 | 80 mg LY2127399 | Placebo
Number analyzed (Participants) | 32 | 26 | 33
Percentage of Lymphocytes | -2.26 (4.651) | -2.20 (4.517) | -0.59 (4.856)
Statistical Analysis 1: Comparison: 30 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA
Statistical Analysis 2: Comparison: 80 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.015, ANCOVA

18. Secondary Outcome: Pharmacodynamics: Change From Baseline in Serum Immunoglobulins at Week 16
Description: Serum immunoglobulin measured by Immunoglobulin A (IgA), Immunoglobulin G (IgG), and Immunoglobulin M (IgM) levels.
Time Frame: Baseline, 16 weeks
Population: Intention to treat (ITT) population defined as participants who were randomized, received at least one dose of study drug, and had at least one post-baseline serum immunoglobulin assessment; last observation carried forward (LOCF). Two participants from sites with good clinical practice [GCP] violations are excluded.
Measure: Mean (Standard Deviation); unit: gram/Liter
Arm/Group | 30 mg LY2127399 | 80 mg LY2127399 | Placebo
Number analyzed (Participants) | 34 | 28 | 35
gram/Liter
  Immunoglobulin G | -0.83 (1.233) | -1.33 (2.055) | -0.62 (1.783)
  Immunoglobulin M | -0.27 (0.325) | -0.24 (0.371) | -0.05 (0.388)
  Immunoglobulin A | -0.24 (0.429) | -0.26 (0.405) | -0.23 (0.729)
Statistical Analysis 1: Comparison: 30 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.146, ANCOVA — p-value is for Immunoglobulin G change at week 16 (LOCF)
Statistical Analysis 2: Comparison: 80 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.125, ANCOVA — p-value is for Immunoglobulin G change at week 16 (LOCF)
Statistical Analysis 3: Comparison: 30 mg LY2127399 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — p-value is for Immunoglobulin M change at week 16 (LOCF)
Statistical Analysis 4: Comparison: 80 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.005, ANCOVA — p-value is for Immunoglobulin M change at week 16 (LOCF)
Statistical Analysis 5: Comparison: 30 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.115, ANCOVA — p-value is for Immunoglobulin A change at week 16 (LOCF)
Statistical Analysis 6: Comparison: 80 mg LY2127399 vs Placebo; Test type: Superiority or Other; p = 0.019, ANCOVA — p-value is for Immunoglobulin A change at week 16 (LOCF)

19. Secondary Outcome: Pharmacokinetics: Predicted Population Mean Parameter: C-trough Steady-state
Description: C-trough is defined as the concentration of LY at the end of the dosing interval at steady state. Mean C-trough value was obtained by conducting a simulation consisting of 1000 participants. The simulated data were then used to determine the noncompartmental PK parameters for each regimen. Mean and standard deviation of the Ctrough values were calculated for each dose group based on simulated data.
Time Frame: Pre-dose, Day 1 through Week 24
Population: All randomized participants with evaluable PK C-trough data.
Measure: Mean (Standard Deviation); unit: Micrograms per Milliliter
Arm/Group | 30 mg LY2127399 | 80 mg LY2127399
Number analyzed (Participants) | 35 | 28
Micrograms per Milliliter | 5.84 (2.87) | 18.9 (7.86)

20. Secondary Outcome: Pharmacokinetics: Predicted Population Mean Parameter: T-half Life (t1/2, Tau)
Description: T-half life (t1/2, tau) is defined as the apparent steady state elimination within the dosing interval. T-half life was obtained by conducting a simulation consisting of 1000 participants using the study drug regimens (30 and 80 mg, intravenous infusion over 30 minutes, once every 3 weeks). The simulated data were then used to determine the noncompartmental PK parameters for each regimen. Mean and standard deviation of the t-half life values were calculated for each dose group based on simulated data.
Time Frame: Pre-dose, Day 1 through Week 24
Population: All randomized participants with evaluable PK t-half life data.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 30 mg LY2127399 | 80 mg LY2127399
Number analyzed (Participants) | 35 | 28
Days | 19 (8) | 22 (8)

ADVERSE EVENTS:
Groups:
- 30 mg LY2127399 - With Rescue Treatment: Participants who were randomized to 30 mg LY2127399 during Treatment Phase who did not have an improvement of at least 20% in either their tender or their swollen joint counts, based on 28 joints at Week 16 assessments and chose to receive optional rescue treatment of an additional 30 minute infusion of 80 mg LY2127399 at Week 16.
- 80 mg LY2127399 - With Rescue Treatment: Participants who were randomized to 80 mg LY2127399 during Treatment Phase who did not have an improvement of at least 20% in either their tender or their swollen joint counts, based on 28 joints at Week 16 assessments and chose to receive optional rescue treatment of an additional 30 minute infusion of 80 mg LY2127399 at Week 16.
- Placebo - With Rescue Treatment: Participants who were randomized to placebo during Treatment Phase who did not have an improvement of at least 20% in either their tender or their swollen joint counts, based on 28 joints at Week 16 assessments and chose to receive optional rescue treatment of an additional 30 minute infusion of 80 mg LY2127399 at Week 16.
- 30 mg LY2127399 - Follow-up: Participants who were randomized to 30 mg LY2127399 during Treatment Phase who required additional follow-up for monitoring of their B cell counts, regardless of whether or not they received optional rescue treatment of an additional 30 minute infusion of 80 mg LY2127399 at Week 16.
- 80 mg LY2127399 - Follow-up: Participants who were randomized to 80 mg LY2127399 during Treatment Phase who required additional follow-up for monitoring of their B cell counts, regardless of whether or not they received optional rescue treatment of an additional 30 minute infusion of 80 mg LY2127399 at Week 16.
- Placebo - Follow-up: Participants who were randomized to placebo during Treatment Phase who required additional follow-up for monitoring of their B cell counts, regardless of whether or not they received optional rescue treatment of an additional 30 minute infusion of 80 mg LY2127399 at Week 16.
Arm/Group | 30 mg LY2127399 - Treatment | 80 mg LY2127399 - Treatment | Placebo - Treatment | 30 mg LY2127399 - Without Rescue Treatment | 30 mg LY2127399 - With Rescue Treatment | 80 mg LY2127399 - Without Rescue Treatment | 80 mg LY2127399 - With Rescue Treatment | Placebo - Without Rescue Treatment | Placebo - With Rescue Treatment | 30 mg LY2127399 - Follow-up | 80 mg LY2127399 - Follow-up | Placebo - Follow-up
Serious Adverse Events (participants affected / at risk) | 1/35 | 2/30 | 3/35 | 0/19 | 1/12 | 0/15 | 0/11 | 0/10 | 0/20 | 0/9 | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 22/35 | 21/30 | 22/35 | 2/19 | 5/12 | 6/15 | 3/11 | 3/10 | 11/20 | 1/9 | 4/11 | 1/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 30 mg LY2127399 - Treatment (N=35) | 80 mg LY2127399 - Treatment (N=30) | Placebo - Treatment (N=35) | 30 mg LY2127399 - Without Rescue Treatment (N=19) | 30 mg LY2127399 - With Rescue Treatment (N=12) | 80 mg LY2127399 - Without Rescue Treatment (N=15) | 80 mg LY2127399 - With Rescue Treatment (N=11) | Placebo - Without Rescue Treatment (N=10) | Placebo - With Rescue Treatment (N=20) | 30 mg LY2127399 - Follow-up (N=9) | 80 mg LY2127399 - Follow-up (N=11) | Placebo - Follow-up (N=10)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 30 mg LY2127399 - Treatment (N=35) | 80 mg LY2127399 - Treatment (N=30) | Placebo - Treatment (N=35) | 30 mg LY2127399 - Without Rescue Treatment (N=19) | 30 mg LY2127399 - With Rescue Treatment (N=12) | 80 mg LY2127399 - Without Rescue Treatment (N=15) | 80 mg LY2127399 - With Rescue Treatment (N=11) | Placebo - Without Rescue Treatment (N=10) | Placebo - With Rescue Treatment (N=20) | 30 mg LY2127399 - Follow-up (N=9) | 80 mg LY2127399 - Follow-up (N=11) | Placebo - Follow-up (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site phlebitis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic mass (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis of male external genital organ (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Granuloma inguinale (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laboratory test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymph node palpable (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 8 (8) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trichorrhexis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ex-tobacco user (Social circumstances) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Poor venous access (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days